CLINICAL TRIAL: NCT00273195
Title: Clinical Investigation of the Medtronic EnTrust™ Implantable Cardioverter Defibrillator (ICD), Model D153ATG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Ventricular Arrhythmias
Keywords: Implantable Cardioverter Defibrillator, Anti-tachycardia pacing (ATP)
MeSH Terms: interventions — Defibrillators, Implantable

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator

SUMMARY:
People who have a dangerously fast heart beat, or whose heart is at risk of stopping beating, may be in need of an electronic device called an implantable cardioverter defibrillator (ICD). An ICD is implanted surgically just under the skin in the upper chest area and it sends a strong electrical impulse, or shock, to the heart to return it to a normal rhythm.

The purpose of this study was to evaluate the safety and efficacy of the EnTrust ICD device. A feature of this device allows it to send small, painless electrical impulses (Anti-tachycardia pacing or ATP) to the heart instead of shocking it out of a rhythm that is too fast. Stopping a dangerous heart rhythm this way does not cause any pain whereas a shock to the heart can feel like a punch in the chest. This device also allows the heart to beat on its own when it can and helping it (by pacing, or sending it electrical signals) when it needs help. This feature is important because previously studies have shown that pacing the heart too often can increase the risk for heart failure or for atrial fibrillation (having too rapid of heart beats in the atrium).

This study is now complete and the device has since been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

Subjects with failure but no symptoms (NYHA Class I) or subjects with mild heart failure that only sometimes interferes with daily activities (NYHA Class II)

Subjects who have, or are risk of having, a heart beat that is too fast and his/her doctor has determined he/she needs an implantable cardioverter defibrillator (ICD)

Subjects who have, or are at risk of developing, rapid beats in the upper chambers of the heart (atrial tachyarrhythmias)

Exclusion Criteria:

Subjects with rapid heart beats in their ventricles (lower chambers of the heart) associated only with reversible causes

Subjects with mechanical tricuspid heart valves (A structure in the heart, located between the right atrium and right ventricle, which allows blood to flow down from the atrium into the ventricle.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-04; Study Completion 2005-06

PRIMARY OUTCOMES:
Safety and efficacy at three months.

SECONDARY OUTCOMES:
To evaluate how well the device distinguished between arrhythmias originating in the atrium versus those that originate in the ventricle.
To evaluate how well the anti-tachycardia pacing function works.
To observe the overall performance of the device system.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (24):
  - Little Rock, Arkansas
  - Glendale, California
  - Inglewood, California
  - Atlantis, Florida
  - Orlando, Florida
  - Macon, Georgia
  - Fort Wayne, Indiana
  - Davenport, Iowa
  - Des Moines, Iowa
  - Salisbury, Maryland
  - Boston, Massachusetts
  - Kansas City, Missouri
  - St Louis, Missouri
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Abington, Pennsylvania
  - Lancaster, Pennsylvania
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Austria (2):
  - Sankt Pölten
  - Steyr
- Canada (6):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Kingston, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Copenhagen, Denmark
- Germany (6):
  - Bonn
  - Göttingen
  - Heidelberg
  - Kaiserslautern
  - München
  - Münster
- Eindhoven, Netherlands
- Basel, Switzerland